CLINICAL TRIAL: NCT06351826
Title: Effectiveness of ELLASI Intervention Towards Response Time, Deterioration, and Metabolic Status of Polytrauma Patients in the Emergency Department
Brief Title: Effectiveness of ELLASI Intervention Towards Polytrauma Patients in the Emergency Department
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Siti Nurlaelah, Effectiveness of ELLASI Intervention Towards Response Time, Deterioration, and Metabolic Status of Polytrauma Patients in the Emergency Department, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22070876
Record Dates: First submitted 2024-01-17; First posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Polytrauma
MeSH Terms: conditions — Multiple Trauma

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ELLASI (Experimental): Polytrauma patients in the intervention group will receive a-6-points structured intervention abbreviated with ELLASI:
  1. Evaluasi: Evaluation of airway and cervical control, remove the foreign body, fluid, etc., from the airway
  2. Letakkan: patient positioning and give oxygen, head-up.
  3. Lakukan: Stabilisasation, including IV insertion, applying pressure and bandage, place monitor, haemodynamic monitoring
  4. Assessment: re-assessment of pain and other main complaints
  5. Siapkan: make sure informed consents are documented
  6. Informasikan: inform patient and family for further intervention
  Interventions: Other: ELLASI
- Standard (Active Comparator): Polytrauma patients in the control group will receive the usual/standard intervention.
  Interventions: Other: Standard

INTERVENTIONS:
Other: ELLASI — A structured intervention for polytrauma patients
  Arms: ELLASI
Other: Standard — Unstructured interventions that are given in everyday practice (standard intervention)
  Arms: Standard

SUMMARY:
This clinical trial aims to test the effectiveness of ELLASI intervention in response time, deterioration score, and metabolic status of polytrauma patients in the emergency department. The main questions it aims to answer are:

1. Is the response time of polytrauma patients who receive ELLASI in the intervention group faster than the control group?
2. Is the deterioration score of polytrauma patients who receive ELLASI in the intervention group better than the control group?
3. Is the metabolic status of polytrauma patients who receive ELLASI in the intervention group better than the control group?

Polytrauma patients in the intervention group will receive ELLASI, a structured intervention consisting of the six following:

1. Evaluation of airway and cervical control, remove the foreign body, fluid, etc., from the airway,
2. Patient positioning and giving oxygen, head-up,
3. Stabilisation, including IV insertion, applying pressure and bandage, place monitor, and haemodynamic monitoring
4. Assessment: re-assessment of pain and other main complaints
5. Make sure informed consents are documented
6. Inform patient and family for further intervention

Polytrauma patients in the control group will receive the usual/standard intervention.

Response time, early warning score, and arterial blood gas of polytrauma patients from both groups will be obtained and documented before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Polytrauma patients
* Have not received medical treatment before

Exclusion Criteria:

* Canceled registration
* Polytrauma patients who are unwilling to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-01-03 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Response time | Immediately before and after the intervention
  Documented from the beginning of ELLASI and standard interventions are delivered to the ending.
Deterioration score | Immediately before the intervention start and 3 hours after the intervention end
  Measured with Early Warning Score system used in the hospital where the data was collected. The scores range from 0 to 14. Higher scores mean deterioration
Acidic Level (pH) | Immediately before the intervention start and 3 hours after the intervention end
  Measure pH of arterial blood gas
Base Excess (BE) | Immediately before the intervention start and 3 hours after the intervention end
  Measure BE of arterial blood gas
Bicarbonate level (HCO3) | Immediately before the intervention start and 3 hours after the intervention end
  Measure HCO3 of arterial blood gas

CONTACTS AND LOCATIONS:
Locations (1):
- RSCM, Jakarta Pusat, West Java, Indonesia

IPD SHARING:
Plan to Share IPD: No
IPD will only be shared with supervisors for consultation. Due to privacy and anonymity, no participants' identifiers that will be disclosed